CLINICAL TRIAL: NCT02206048
Title: Use of High-Resolution Microendoscopy (HRME) in Patients With Adenocarcinoma In-Situ (AIS) of the Cervix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-0885; 14037870 (Other: Institution of Medicine (IOM)); NCI-2014-01790 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Results first posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Cervix Carcinoma
Keywords: Cervix Carcinoma; Cervical adenocarcinoma in situ; AIS; Cervical intraepithelial neoplasia; CIN; microinvasive carcinoma of the cervix; cold knife cone of the cervix; CKC; High-Resolution Microendoscopy; HRME; Proflavine
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia | interventions — Proflavine; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- High-Resolution Microendoscopy (HRME) (Experimental): Before participant's cold knife cone biopsy (CKC), topical application of 0.01% proflavine solution applied to cervix. HRME probe applied to cervix and high-resolution images obtained. Participant undergoes cervical biopsies of any abnormal areas noted with colposcopy and/or HRME. Immediately following the CKC, the removed surgical specimen evaluated. Proflavine reapplied to surgical specimen and repeat evaluation with HRME performed and high-resolution images obtained.
  Interventions: Drug: Proflavine; Procedure: High-Resolution Microendoscopy (HRME) Imaging

INTERVENTIONS:
Drug: Proflavine — 0.01% proflavine solution topically applied to cervix before high-resolution microendoscopy (HRME) imaging.
Procedure: High-Resolution Microendoscopy (HRME) Imaging — in-vivo high-resolution microendoscopy (HRME) images of cervical adenocarcinoma in situ (AIS) performed immediately prior to conization.
  Other Names: HRME

SUMMARY:
The goal of this clinical research study is to learn if it is possible to get high-resolution microendoscopy (HRME) images of AIS tissue and/or tissue from microinvasive carcinoma right before a biopsy of the cervix. Researchers also want to learn if HRME images can show the difference between cancerous tissue and normal cervical tissue.

DETAILED DESCRIPTION:
If you agree to take part in this study, after you are in the operating room and under general anesthesia, proflavine hemisulfate solution (contrast dye) will be applied to the cervix. Images will be collected with the probe from the HRME device. The HRME probe is a long thin tube with a camera at the tip. This probe will be applied to the cervix and images obtained. These images will be used for research. This should add about 10 minutes to the total time you are in the operating room.

There will be no change to the planned standard-of-care colposcopy and biopsy.

Follow-Up:

A member of the research team will call you within 30 days after the procedure to ask how you are feeling and if you are having any symptoms. This call should last about 5 minutes.

Length of Study:

Your active participation in this study will be over after the biopsy.

This is an investigational study. The goal of this clinical research study is to learn if it is possible to get high-resolution microendoscopy (HRME) images of AIS tissue and/or tissue from microinvasive carcinoma right before a biopsy of the cervix. Researchers also want to learn if HRME images can show the difference between cancerous tissue and normal cervical tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Any woman with a confirmed preoperative diagnosis of cervical AIS, including co-existing squamous CIN and/or microinvasive cancer
2. Women undergoing cold knife cone (CKC) of the cervix at MD Anderson
3. Negative pregnancy test for women of child-bearing potential
4. Women who are >/= 21 years of age and < 65 years of age
5. Ability to understand and the willingness to provide informed consent and sign a written Informed Consent Document (ICD)

Exclusion Criteria:

1. Women < 21 years of age and >/= 65 years of age
2. Women with a known allergy to proflavine or acriflavine
3. Women who are pregnant or nursing
4. Patients unable or unwilling to provide informed consent or sign a written Informed Consent Document (ICD)

Ages: 21 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2015-10-02 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Schmeler, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High-Resolution Microendoscopy (HRME)
Started | 9
Completed | 8
Not Completed | 1
Not completed — Change in OR schedule and availability of study staff | 1

BASELINE CHARACTERISTICS:
Arm/Group | High-Resolution Microendoscopy (HRME)
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Acquiring In-vivo High-Resolution Microendoscopy (HRME) Images of Cervix Prior to Conization
Description: Methodology determined feasible if in-vivo HRME images are acquired in if 18 of the 20 participants enrolled in the study.
Time Frame: 1 day
Population: Due to not meeting enrollment requirements, data was not collected
Arm/Group | High-Resolution Microendoscopy (HRME)
Number analyzed (Participants) | 0

2. Secondary Outcome: Adenocarcinoma In-Situ (AIS) Distinguished From Normal Cervical Tissue Using High-Resolution Microendoscopy (HRME) Imaging
Description: AIS finding tabulated by the CKC specimen results as determined by pathology. Concordance of HRME images taken ex-vivo estimated with pathology findings with a 90% credible, assuming a beta (1.8, 0.2) prior distribution for the concordance.
Time Frame: 1 day
Population: Due to low accrual, no specimens were collected to be analyzed
Arm/Group | High-Resolution Microendoscopy (HRME)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events will be captured from the time of the first protocol-specific intervention, until 30 days after the last dose of drug, unless the participant withdraws consent. Serious adverse events must be followed until clinical recovery is complete and laboratory tests have returned to baseline, progression of the event has stabilized, or there has been acceptable resolution of the event.
Arm/Group | High-Resolution Microendoscopy (HRME)
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
Due to low accrual no analysis conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT02206048/Prot_SAP_000.pdf